CLINICAL TRIAL: NCT06823843
Title: The Effect of Sublingual Nitroglycerin on Absolute Coronary Blood Flow: A Randomised, Placebo-controlled, Mechanistic Trial
Brief Title: The Effect of Sublingual Nitroglycerin on Absolute Coronary Blood Flow
Acronym: FLOW-NITRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VZW Cardiovascular Research Center Aalst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OLV2024/037; B1262024000004
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Coronary Arterial Disease (CAD); Angina (Stable)
Keywords: nitroglycerin (GTN); angina; coronary artery disease; absolute coronary flow; continuous intracoronary thermodilution
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Coronary Artery Disease | interventions — Nitroglycerin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 2 puffs of sublingual saline
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)
- GTN (Experimental): 2 puffs for a total dose of 800 µg
  Interventions: Drug: Glycerin trinitrate (GTN)

INTERVENTIONS:
Drug: Glycerin trinitrate (GTN) — 2 sublingual puffs for a total dose of 800 µg
  Arms: GTN
Drug: Saline (NaCl 0,9 %) (placebo) — 2 puffs of sublingual saline
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effect of sublingual nitroglycerin on absolute coronary blood flow in adult patients undergoing coronary angiography. The main questions it aims to answer are:

* Does sublingual nitroglycerin change absolute coronary blood flow compared to placebo?
* What is the effect of sublingual nitroglycerin on important cardioavascular parameters such as coronary pressure and resistance?

Researchers will compare the sublingual nitroglycerin group to the placebo group to see if nitroglycerin leads to significant changes in coronary blood flow and microvascular function.

Participants will:

* Receive either sublingual nitroglycerin or a placebo during coronary angiography.
* Undergo coronary blood flow measurements before and after the intervention using standardized assessment techniques.

DETAILED DESCRIPTION:
INTRODUCTION

Nitrates remain a key drug class in the management of angina pectoris due to their capacity to decrease myocardial oxygen demand. Their principle mechanism of action relates to the relaxation of vascular smooth muscle leading to vasodilation. Nitrates are predominately venodilators resulting in a decrease in cardiac preload, left ventricular diastolic pressure, and thus myocardial wall stress and subendocardial compression. However, at low doses, nitrates also trigger arterial and arteriolar dilatation with an eventual reduction in systemic vascular resistance and cardiac afterload at higher doses.

At the coronary level, the direct action of nitrates is thought to be almost exclusively restricted to the epicardial vessels with significant vasodilatation demonstrated in both normal and stenotic epicardial coronary arteries. Furthermore, in a canine model, nitrates have been shown to increase absolute coronary blood. The limited direct effect of nitrates on coronary microcirculation relates to the resistance of arterioles with a diameter <100 μm to their action. However, coronary flow in these smaller vessels may be increased indirectly as decreased left ventricular end-diastolic pressure and wall stress induced by systemic venous dilatation has been shown to increase flow from the epicardium to endocardium.

Despite our understanding of the mechanisms behind the antianginal effects of nitrates, the quantification of their effect on absolute coronary flow has never been demonstrated in humans.

GOAL OF THE STUDY

In the present study, the investigators aim to use continuous thermodilution to asses the impact of sublingual nitroglycerin (NTG) on absolute coronary blood flow when compared with a placebo control.

DESIGN

This is an investigator-initiated, prospective, double-blinded randomised controlled study recruiting patients undergoing diagnostic coronary angiography for suspected angina pectoris from a single centre, and in whom coronary blood flow measurements are part of routine clinical practice, patients will be randomised between sublingual NTG and placebo.

OVERVIEW OF THE STUDY PROTOCOL

Critically, all recruited patients will have any pre-existing vasoactive medications stopped 24 hours before the protocol.

Upon completion of diagnostic coronary angiography, baseline and hyperemic, coronary pressures (Pd and Pa) and resting volumetric blood flow (Qrest) will be assessed by continuous thermodilution. These measurements necessitate the use of a pressure/temperature guidewire and a dedicated infusion catheter. They are performed routinely to evaluate the function of the microcirculation. The measurements are described in details hereunder (see paragraph 'Continuous thermodilution measurements').

During the measurement of resting flow, the patient will be randomised to either the intervention (2 puffs of sublingual NTG at a total dose of 800 µg) or a sublingual placebo by a research nurse. The research nurse will administer the sublingual spray with both the physicians and the patient blinded to patient randomisation. Once administered, continuous thermodilution will be continued for a further 7 minutes to permit enough time to capture any treatment effect as seen in the canine model. It is expected that the protocol, including recording of baseline values, will last ~10 minutes. The same protocol will then be repeated during hyperaemia.

The following parameters will be recorded/calculated at baseline as well as at 1, 3, 5, and 7 minutes post NTG administration, in order to capture the full effect of NTG on both coronary and systemic haemodynamics.

* Absolute coronary blood flow (Q)
* Microvascular resistance (Rµ)
* Epicardial resistance (Repi)
* Total resistance (Rtot)
* Aortic pressure (Pa)
* Distal coronary pressure (Pd)

ELIGIBILITY:
Inclusion Criteria:

* Referred for invasive coronary angiography (ICA) for suspected coronary artery disease

Exclusion Criteria:

* ≥1 severe stenosis (defined as a diameter stenosis >70%)
* Clinical signs or symptoms of congestive heart failure
* Severe valvular heart disease requiring either surgical or percutaneous intervention
* History of coronary artery bypass grafting
* Tortuous coronary anatomy in which wire manipulation could be complex
* Significant arrhythmia
* Use of vasoactive medications within 24 hours of coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the absolute coronary flow 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Absolute coronary flow will be measured using continuous intracoronary thermodilution

SECONDARY OUTCOMES:
Change from baseline in the absolute microvascular resistance 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Absolute microvascular resistance will be calculated using absolute coronary flow and distal coronary pressure
Change from baseline in the absolute epicardial resistance 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Absolute epicardial resistance will be calculated using absolute coronary flow, aortic pressure and distal coronary pressure
Change from baseline in aortic pressure 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Aortic pressure will be measured using the coronary guiding catheter
Change from baseline in distal coronary pressure 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Distal coronary pressure will be measured using a standard coronary pressure wire
Change from baseline in left ventricular end-diastolic pressure 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  LVEDP will be measured using a pigtail catheter at baseline, and at the end of the protocol
Change from baseline in left ventricular work 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Left ventricular work will be estimated using the systolic pressure-time index (SPTI) derived from the aortic pressure curve.
Change from baseline in myocardial perfusion 10 minutes after administration of the intervention | 10 minutes from the administration of the sublingual intervention
  Myocardial perfusion will be estimated using the Buckberg Index. It will be calculated by dividing the diastolic pressure-time index (i.e. time of coronary perfusion) by the systolic pressure-time index (i.e. time of myocardial oxygen demand).

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Cardiovascular Center Aalst, Aalst, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
This was included in the original ethical committee sumission